CLINICAL TRIAL: NCT01066858
Title: Maternal and Infant Monitoring for Evidence of Toxicity Related to Tenofovir Exposure: The Bone and Kidney Health Substudy of the IMPAACT 1077 PROMISE Protocol (Promoting Maternal and Infant Survival Everywhere)
Brief Title: Study of Effects of Tenofovir on Bone Health and Kidneys During Pregnancy and Breastfeeding
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Gilead Sciences (Industry)
Responsible Party: Sponsor
Other Study IDs: P1084s (PROMISE); 10790 (Registry Identifier: DAIDS ES); IMPAACT P1084s
Record Dates: First submitted 2010-02-09; First posted 2010-02-10 (Estimated); Last update posted 2022-09-23 (Actual); Status verified 2022-09

CONDITIONS: HIV Infections
Keywords: tenofovir; renal and bone toxicity; pregnancy; breastfeeding; mother to child transmission
MeSH Terms: conditions — HIV Infections; Breast Feeding | interventions — Tenofovir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Maternal/infant antepartum exposure: * HIV-infected women exposed to TDF during pregnancy
  * Infants of HIV-infected women exposed to TDF during pregnancy
  Interventions: Drug: Tenofovir disoproxil fumarate (TDF)
- Maternal/infant postpartum exposure: * HIV-infected women exposed to TDF while breastfeeding
  * Infants of HIV-infected women exposed to TDF while breastfeeding
  Interventions: Drug: Tenofovir disoproxil fumarate (TDF)
- Maternal/infant antepartum no exposure: * HIV-infected women not exposed to TDF during pregnancy
  * Infants of HIV-infected women not exposed to TDF during pregnancy
- Maternal/infant postpartum no exposure: * HIV-infected women not exposed to TDF during breastfeeding
  * Infants of HIV-infected women not exposed to TDF during breastfeeding

INTERVENTIONS:
Drug: Tenofovir disoproxil fumarate (TDF) — Some participants will receive varying doses of TDF during pregnancy or breastfeeding as part of the larger study (IMPAACT 1077 PROMISE).
  Groups: Maternal/infant antepartum exposure; Maternal/infant postpartum exposure

SUMMARY:
The purpose of this study is to look at the effects of tenofovir disoproxil fumarate (an anti-HIV medication) on the bone health and kidneys of women with HIV during pregnancy and while breastfeeding. The study will also look at the changes in overall health, bone health and how the kidneys work in the infants of these women.

DETAILED DESCRIPTION:
A small number of adults (who are not pregnant) and children who take anti-HIV medications develop problems with their kidneys and with the strength of their bones. These problems may be more common when tenofovir disoproxil fumarate (TDF) is used. Studies about these bone and kidney effects have not been done in pregnant and breastfeeding women and their infants.

This is a substudy of a larger study (IMPAACT 1077 PROMISE [Promoting Maternal and Infant Survival Everywhere]) to evaluate the safety of anti-HIV medications used in pregnancy and during breastfeeding. Only participants in the larger study randomly assigned to receive maternal tenofovir disoproxil fumarate (TDF) or no maternal TDF during pregnancy or during breastfeeding will be enrolled in this substudy.

This substudy will look at two groups of participants:

* An antepartum exposure group to look at the effects of TDF during pregnancy
* A postpartum exposure group to look at the effects of TDF during breastfeeding

All mother-infant pairs in the substudy will be followed for 74 weeks after delivery. During this time, the women and their infants will have medical checkups and tests. The tests will include tests of blood, urine, cord blood, and breast milk. Some of the women and infants will have a special x-ray called a dual energy e-ray absorptiometry (DXA) scan to measure bone strength. The timing of the tests-at enrollment, at delivery, at 6, 10, 26, or 74 weeks-will vary dependent on which part of this substudy women and infants are enrolled in. Those in charge of the substudy will try to schedule medical visits and tests at the same time as tests scheduled for the larger IMPAACT 1077 study.

ELIGIBILITY:
Antepartum (AP) Part of Study (TDF Exposure During Pregnancy)

Inclusion Criteria:

* Mother-infant pair enrolled in 1077BA or 1077FA
* At a clinical site that has been approved as a P1084s DXA site
* Enrolled in the substudy up to the Week 2 visit of 1077BA/1077FA (within 21 days after 1077BA/1077FA study entry) and prior to the start of labor
* Willing and able to provide written informed consent to participate in this substudy

Exclusion Criteria:

* None

Postpartum (PP) Part of Substudy (TDF Exposure During Breastfeeding) (Note: this applies only to the new enrollment to P1084s, i.e., those who were not enrolled to P1084s while on the AP component)

Inclusion Criteria:

* Mother and their infant enrolled in 1077BP
* At a clinical site that has been approved as a P1084s DXA site
* Enrolled in the substudy within 6 to 14 days of delivery, on the same day as enrollment in 1077BP
* Willing and able to provide written informed consent to participate in this substudy

Exclusion Criteria:

* TDF exposure during pregnancy [NOTE: TDF use for up to 12 days beginning at labor allowed]
* Enrolled in the AP part of P1084s

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: For antepartum (AP) exposure part of P1084s: Mother/infant pairs enrolled in the antepartum components of 1077BF or 1077FF (1077BA and 1077FA respectively) at African clinical sites approved as P1084s DXA sites.
  For postpartum (PP) exposure part of P1084s: Mothers and their infants enrolled in the postpartum component of 1077BF (107BP) at African clinical sites approved as P1084s DXA sites.
Sampling Method: Non-Probability Sample
Enrollment: 1765 (Actual)
Dates: Start 2011-03-22 (Actual); Primary Completion 2015-11-30 (Actual); Study Completion 2015-11-30 (Actual)

PRIMARY OUTCOMES:
Antepartum Component: Creatinine clearance (CrCl) | For women and infants: at delivery/birth, up to Week 1
  Antepartum Component: Creatinine clearance (CrCl)
Antepartum Component: Bone resorption (Dpyr) | For women and infants: at delivery/birth, up to Week 1
  Antepartum Component: Bone resorption (Dpyr)
Antepartum Component: Lumbar spine bone mineral density (BMD) via dual energy e-ray absorptiometry (DXA) | For women: at delivery/birth, up to Week 1
  Antepartum Component: Lumbar spine bone mineral density (BMD) via dual energy e-ray absorptiometry (DXA)
Antepartum Component: Lumbar spine bone mineral content (BMC) and whole body BMC via DXA | For infants: at delivery/birth, up to Week 1
  Antepartum Component: Lumbar spine bone mineral content (BMC) and whole body BMC via DXA
Antepartum Component: Length-for-age Z-score | For infants: at delivery/birth, up to Week 1 and Week 26
  Antepartum Component: Length-for-age Z-score
Postpartum Component: CrCl | For women: at postpartum entry (delivery/birth, up to Week 1) and Week 74; for infants: at Week 26
  Postpartum Component: CrCl
Postpartum Component: Dpyr | For women: at Week 74; for infants: at Week 26
  Postpartum Component: Dpyr
Postpartum Component: Lumbar spine BMD via DXA | For women: at postpartum entry (delivery/birth, up to Week 1) and Week 74
  Postpartum Component: Lumbar spine BMD via DXA
Postpartum Component: Lumbar spine BMC via DXA | For infants: at Week 26
  Postpartum Component: Lumbar spine BMC via DXA
Postpartum Component: Length-for-age Z-score | For infants: at postpartum entry (delivery/birth, up to Week 1) and Week 26
  Postpartum Component: Length-for-age Z-score

SECONDARY OUTCOMES:
CrCl | For women: Weeks 6, 26, and 74; for infants: at Weeks 10, 26, and 74
  CrCl
BMD | For women: at delivery and change in hip BMD from delivery to Week 74
  BMD
Dpyr | For women: at Weeks 6, 26, and 74; for infants: at Weeks 10, 26, and 74
  Dpyr
Mineral composition of breast milk | For women: at Weeks 1, 6, 26, and 74
  Mineral composition of breast milk
Lumbar spine BMC | For infants: Week 26
  Lumbar spine BMC
Infant growth | For infants: at Weeks 10 and 74
  Infant growth
Concentration of hormonal growth factors (for infants) | For infants: at birth and Weeks 10, 26, and 74
  Concentration of hormonal growth factors (for infants)

CONTACTS AND LOCATIONS:
Overall Officials: George K. Siberry, MD, MPH, Study Chair — NICHD/NIH; Lynda Stranix-Chibanda, MBChB, MMED, Study Chair — University of Zimbabwe
Locations (11):
- Malawi (2):
  - Blantyre CRS, Blantyre
  - Malawi CRS, Lilongwe
- South Africa (5):
  - Soweto IMPAACT CRS, Johannesburg, Gauteng
  - Shandukani Research CRS, Johannesburg, Gauteng
  - Durban Paediatric HIV CRS, Durban, KwaZulu-Natal
  - Umlazi CRS, Durban, KwaZulu-Natal
  - Family Clinical Research Unit (FAM-CRU) CRS, Tygerberg, Western Cape
- MU-JHU Research Collaboration (MUJHU CARE LTD) CRS, Kampala, Mpigi, Uganda
- Zimbabwe (3):
  - Seke North CRS, Chitungwiza
  - St Mary's CRS, Chitungwiza
  - Harare Family Care CRS, Harare

REFERENCES:
- [Background] Foster C, Lyall H, Olmscheid B, Pearce G, Zhang S, Gibb DM. Tenofovir disoproxil fumarate in pregnancy and prevention of mother-to-child transmission of HIV-1: is it time to move on from zidovudine? HIV Med. 2009 Aug;10(7):397-406. doi: 10.1111/j.1468-1293.2009.00709.x. Epub 2009 May 12. PMID 19459986
- [Background] Nurutdinova D, Onen NF, Hayes E, Mondy K, Overton ET. Adverse effects of tenofovir use in HIV-infected pregnant women and their infants. Ann Pharmacother. 2008 Nov;42(11):1581-5. doi: 10.1345/aph.1L083. Epub 2008 Oct 28. PMID 18957630
- [Derived] Baltrusaitis K, Makanani B, Tierney C, Fowler MG, Moodley D, Theron G, Nyakudya LH, Tomu M, Fairlie L, George K, Heckman B, Knowles K, Browning R, Siberry GK, Taha TE, Stranix-Chibanda L; PROMISE P1084s Study Team. Maternal and infant renal safety following tenofovir disoproxil fumarate exposure during pregnancy in a randomized control trial. BMC Infect Dis. 2022 Jul 20;22(1):634. doi: 10.1186/s12879-022-07608-8. PMID 35858874
- [Derived] Stranix-Chibanda L, Tierney C, Sebikari D, Aizire J, Dadabhai S, Zanga A, Mukwasi-Kahari C, Vhembo T, Violari A, Theron G, Moodley D, George K, Fan B, Sommer MJ, Browning R, Mofenson LM, Shepherd J, Nelson B, Fowler MG, Siberry GK; PROMISE P1084s study team. Impact of postpartum tenofovir-based antiretroviral therapy on bone mineral density in breastfeeding women with HIV enrolled in a randomized clinical trial. PLoS One. 2021 Feb 5;16(2):e0246272. doi: 10.1371/journal.pone.0246272. eCollection 2021. PMID 33544759